CLINICAL TRIAL: NCT04205760
Title: Preoperative Nutritional Optimization and Physical Exercise for Patients Scheduled for Elective Implantation for a Left-Ventricular Assist Device
Acronym: PROPER-LVAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Christian Stoppe, Prof. Dr. med., RWTH Aachen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-136
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Left Ventricular Assist Device; End-stage Heart Failure; Cardiac Surgery
Keywords: LVAD; preoperative optimization; end-stage heart failure; cardiac surgery; nutrition therapy; exercise; cycling
MeSH Terms: conditions — Motor Activity | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Intervention Model Description: National multicenter two-group randomized-controlled, blinded to assessor clinical pilot trial
Who Masked: Outcomes Assessor
Masking Description: functional outcome assessor will be blinded to study group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard Care as per local guidelines
- Intervention (Experimental): Oral nutrition support (ONS) and bed-cycling before surgery
  Interventions: Combination Product: Nutrition + exercise

INTERVENTIONS:
Combination Product: Nutrition + exercise — Patients will receive preoperative optimization consisting of oral nutrition support (Fresubin 3.2 kcal) and bed-cycling (50 minutes per day) for 5-14 days before surgery.
  Other Names: bed cycling; ONS
  Arms: Intervention

SUMMARY:
This is a pilot, randomized, multicenter interventional trial of a combined preoperative oral nutritional support (ONS) and physical exercise therapy in patients planned for elective implantation of a left-ventricular assist device (LVAD). This pilot study pursues to demonstrate the feasibility and safety of a study protocol to optimize the patients' nutritional and physical state to reduce the number of postoperative complications and consequently to ameliorate the patients' outcome.

DETAILED DESCRIPTION:
The oral nutrition supplementation will be started immediately after randomization and will be continued until surgery. The patients will receive a dosage of ONS adjusted to their nutritional risk. Regular monitoring of blood sugars, electrolytes, phosphate, and triglycerides will occur twice per week, as per standard protocol.

In-bed cycling will be started as soon as possible after randomization. Cycling sessions will be performed daily for 50 minutes, at least 5 times a week until surgery. Standard safety criteria will be assessed prior to initiating cycling treatments. The in-bed cycling will be performed passively or actively with graded increasing resistance. All cycling interventions will be performed under 1:1 supervision of medically trained study personnel while monitoring patient's heart rate, systolic and diastolic blood pressure and transcutaneous oxygen saturation of blood.

When evaluating the effect of a combined nutritional and exercise intervention, other important co-interventions should be standardized to reduce potential confounding of trial outcomes. All study patients should be fed with an oral diet that is in accordance to local standards, whereas it is strongly recommended to adhere to current clinical practice guidelines. Besides, the investigators highly encourage daily respiratory therapy in both groups plus mobilization as much as feasible.

All other key interventions during preoperative treatment will be standardized in accordance to the local clinical practice. Study teams will follow up on the patients on a daily base, documenting adherence with study interventions and key co-interventions.

Patients in the control group will not receive preoperative ONS. No bed cycling will be allowed from admission until surgery. Neither of these practices are the current standard of care in the participating unit.

ELIGIBILITY:
Inclusion Criteria:

1. Given informed consent
2. Adult patients (≥18 years)
3. Patients undergoing elective LVAD implantation Additional cardiac surgery, such as bypass grafting, or valve repair is permitted

Exclusion Criteria:

1. Hospital admission <5 days prior to planned LVAD implantation
2. Patients on ECMO or INTERMACS<1
3. Patients already receiving nutrition support on hospital admission
4. Enteral nutrition is contraindicated.
5. Pregnant or lactating patients
6. Patients with clinical fulminant hepatic failure
7. Patients with cirrhosis Child's Class C Liver Disease
8. Patients with clinical kidney failure or requiring hemodialysis
9. Known allergy or intolerance to study nutrients
10. Intracranial or spinal process affecting motor function
11. Lower extremity impairments that prevent cycling
12. Disabling neuropsychiatric disorders or language barriers
13. Weight > 150 kg
14. Enrolment in an industry sponsored randomized trial within the last 30 days (co-enrolment in academic randomized trials will be considered on a case by case basis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-07-02 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of adverse events | up to 2 weeks before surgery
  adverse events between groups related to cycling and nutritional complications
Separation of caloric supplementation | up to 2 weeks before surgery
  Separation between groups on prescribed caloric targets
Separation of protein supplementation | up to 2 weeks before surgery
  Separation between groups on prescribed protein targets
Proportion of interventions received as prescribed | up to 2 weeks before surgery
  Proportion of interventions received as prescribed
Rate of patients recruited per month | up to 18 months
  Target: 1.5 patients per month
Ratio of control patients received physiotherapy | up to 2 weeks before surgery
  Ratio of control patients received physiotherapy
Ratio of control patients received nutritional support | up to 2 weeks before surgery
  Ratio of control patients received nutritional support

SECONDARY OUTCOMES:
mortality rates at day 30 | day 30 after randomization
  mortality rates at day 30
rates of ICU length of stay | up to 3 months
  rates of ICU length of stay
rates of hospital length of stay | up to 3 months
  rates of hospital length of stay
Mean duration of mechanical ventilation | up to 3 months
  Mean duration of mechanical ventilation
Incidence of complications | up to 3 months
  Incidence of complications
Incidence of infections | up to 3 months
  Incidence of infections
Change in Mid-arm circumference | up to 6 months
  baseline values versus follow-up values
Change in Muscle mass - Quadriceps thickness | up to 6 months
  ultrasound, baseline values versus follow-up values
Change in Muscle mass - Quadriceps cross sectional area | up to 6 months
  ultrasound, baseline values versus follow-up values
Change in Muscle strength - Handgrip strength | up to 6 months
  Dynamometry, baseline values versus follow-up values
Change in Muscle strength - Quadriceps strength | up to 6 months
  Dynamometry, baseline values versus follow-up values
Change of Clinical Frailty score (CFS) | up to 6 months
  baseline values versus follow-up values; Score: 1-9 (very fit: 1, terminally ill: 9)
Change in Physical function - 6-Minute Walk Test | up to 6 months
  baseline values versus follow-up values, 6-minute walking distance
Change in Physical function - Short Physical Performance Battery | up to 6 months
  baseline values versus follow-up values,(Score: 0-12; 0=worst performance and 12=best performance)
Change in Physical function - Functional Status Score for the ICU | up to 6 months
  baseline values versus follow-up values,(Score 0-35; the higher the score, the better physical functioning)
Change in quality of life - Lawton Instrumental Activities of Daily Living (IADL) | up to 6 months
  baseline values versus follow-up values, (score 0-8; the higher the more independent)
Change in quality of life - Katz Activities of Daily Living (ADL) | up to 6 months
  baseline values versus follow-up values,(Score: 0-100; the higher the more independent)
Quality of life - Short Form 36 (SF-36) | up to 6 months
  baseline values versus follow-up values,(Score: 0-100; 100=no limitation in daily life and 0=completely limited)
Change in neurological function - Mini Mental State Examination | up to 6 months
  baseline values versus follow-up values, (score: 0-30; the higher the less cognitively impaired)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Stoppe, Prof. Dr. med., Principal Investigator — RWTH Aachen University
Locations (5):
- Germany (5):
  - Heart Center Bad Oeynhausen, Bad Oeynhausen, North Rhine-Westphalia
  - RWTH Aachen University, Aachen
  - Heart Center Dresden, Dresden
  - University Hospital Justus-Liebig University Giessen, Giessen
  - University Medical Center Schleswig-Holstein, Campus Kiel, Kiel

IPD SHARING:
Plan to Share IPD: Undecided